CLINICAL TRIAL: NCT06524141
Title: A Review of the Current Situation in Following Difficult Airway Guidelines: a Survey
Brief Title: Review of the Follow-up of Difficult Airway Guidelines
Status: Active, not recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-47
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia; Airway Management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This questionnaire study aimed to ask the participants selected questions from the recommendations of the main guidelines on airway management. Thus, the compliance rate of anesthesiologists with the guidelines in different difficult airway management situations will be investigated. Secondarily, it was aimed to raise awareness about the recommendations of the guidelines.

ELIGIBILITY:
Inclusion Criteria:

* To be a specialist in Anesthesiology and Reanimation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians who have completed Anesthesiology and Reanimation specialty training
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Anesthesiologists' adherence to current guidelines in difficult airway management situations. | 5 months
  The study aims to ask the participants questions selected from the recommendations of the main guidelines on airway management. The compliance rate of anesthesiologists with guidelines in difficult airway management situations will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli City Hospital, Kocaeli, Turkey (Türkiye)